CLINICAL TRIAL: NCT03622372
Title: Pivotal, Randomised, Controlled Trial to Evaluate the Safety and Effectiveness of the CoNextions TR Implant System for Zone 2 Flexor Tendon Repair
Brief Title: Zone 2 Flexor Tendon Repair With CoNextions TR Implant System
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CoNextions Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRFDP1
Record Dates: First submitted 2018-07-18; First posted 2018-08-09 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Tendon Injury - Hand
Keywords: FLEXOR TENDON; ZONE 2

STUDY DESIGN:
Intervention Model Description: Participants will be assigned using a 1:1 randomization scheme to receive either the investigational device or a suture repair for the surgical treatment of their tendon lacerations.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and the Occupational Therapist performing the majority of the outcome assessments will be masked to the treatment until the 12 week post-operative visit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- CoNextions TR Implant (Experimental): Operative repair of Zone 2 FDP tendon lacerations will be performed using the CoNextions TR Implant System
  Interventions: Procedure: Operative repair of Zone 2 FDP tendon lacerations; Device: CoNextions TR Implant System
- Suture Repair (Active Comparator): Operative repair of Zone 2 FDP tendon lacerations will be performed using a 4-strand locked cruciate repair utilizing either 3.0 or 4.0 prolene suture
  Interventions: Procedure: Operative repair of Zone 2 FDP tendon lacerations; Device: 4-strand locked cruciate repair

INTERVENTIONS:
Procedure: Operative repair of Zone 2 FDP tendon lacerations — Zone 2 tendon laceration(s) will be surgically repaired either using the experimental device or the active comparator
Device: CoNextions TR Implant System — The CoNextions TR Implant System will be used to repair Zone 2 FDP tendon laceration(s).
  Arms: CoNextions TR Implant
Device: 4-strand locked cruciate repair — A 4-strand locked cruciate repair utilizing either 3.0 or 4.0 prolene suture will be used to repair Zone 2 FDP tendon laceration(s).
  Arms: Suture Repair

SUMMARY:
Prospective, randomised, controlled trial of a novel implant intended for use during surgical repair of lacerated Zone 2 flexor digitorum profundus tendons.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Willing and able to provide a signed and dated informed consent form
3. Stated willingness to comply with all study procedures
4. Available for the duration of the study
5. Have one or two fully lacerated digital FDP tendon(s), with or without a concomitant injury of the flexor digitorum superficialis, in Zone 2 of the index, middle, ring, or small finger
6. Tendon laceration occurred within the previous 14 days

Exclusion Criteria:

1. Pregnant or planning to become pregnant during the follow-up period
2. Autoimmune disorder(s)
3. Type 1 diabetes mellitus or clinical history of poorly controlled Type 2 diabetes mellitus
4. Lack of proper cutaneous coverage at repair site
5. Concomitant fracture
6. Amputated digit(s)
7. Arthritis of the hand
8. Prior hand trauma with residual impact to function
9. Congenital hand defect
10. Conditions that would affect comparative measurements in the uninjured hand
11. Tendon laceration caused by a crush injury
12. Prior sensory impairment in digits of either hand. Note: Participants with nerve injuries associated with the trauma causing the current flexor tendon injury are eligible for enrollment
13. Vascular injuries that require revascularisation procedures
14. Ischemia and/or blood supply compromise
15. Prior or current infections at or near the intended implant site
16. Active sepsis, MRSA, or other conditions that may prevent healing
17. History of foreign-body sensitivity to 316 L Stainless Steel or UHMWPE
18. Implantation of CoNextionsTR Implant would result in physical contact with other metal implants made of material other than implant grade stainless steel such as titanium, titanium alloys, cobalt chromium, or other dissimilar metals
19. Any condition(s) which, in the opinion of the investigator, may impact the participant's ability to properly follow-up or otherwise be at-risk for following protocol instructions
20. Currently participating in another clinical/device trial

    The following criteria, determined during the surgical procedure, will also cause an individual to be excluded from the study:
21. Surgical site access less than 20 mm in total or less than 10 mm on either side of intended implant site
22. Injured tendon is outside of the width range (3.0-7.0 mm) and thickness range (1.5-4.0 mm) specified for the CoNextionsTR Implant System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate of tendon re-rupture | 24 weeks
  Primary Safety Endpoint
Mobility of the affected digits using Strickland's Revised Score | 24 weeks
  Primary Effectiveness Endpoint-Strickland's Revised Score provides a descriptive measure of the mobility of digits. Range of motion measurements taken on the studied digits are used to generate a score on a 0 (least mobile) to 100 (most mobile) with outcomes being classified as: excellent (75-100%), good (50-784%), fair (25-49%), or poor (<25%).

SECONDARY OUTCOMES:
Visual Analog Score (VAS) for Pain Assessment (0-10 cm scale) | 24 weeks
  Patient reported pain intensity measuring from 0 (no pain) to 10 (worst imaginable pain).
Surgical Site Infection | 24 weeks
  Presence of infection at the surgical site
Disabilities of the Arm, Shoulder and Hand Questionnaire (DASH) Questionnaire | 24 weeks
  DASH is a patient-reported questionnaire consisting of 30 questions designed to evaluate a patients ability to perform certain upper extremity activities. The patients answers are used to calculate a score from 1 (most disabled) to 100 (least disabled). DASH is validated to be able to detect small and large changes over time, most notably before and after surgical interventions in the upper extremity.
Grip Strength measured using a dynamometer with values for the affected hand being calculated as a percentage of the grip strength of the unaffected hand | 24 weeks
  The average of three grip strength values taken in succession (kilograms).
Tip pinch strength measured with a pinch gauge with values for the affected fingers calculated as a percentage of the tip pinch strength for corresponding fingers on the unaffected hand | 24 weeks
  The average of three tip pinch strength values taken in succession (kilograms).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Solomons, MD, Principal Investigator — Grootte Schuur Hospital
Locations (4):
- South Africa (4):
  - Grootte Schuur Hospital, Cape Town
  - Tygerberg Hospital, Cape Town
  - Inkosi Albert Luthuli Central Hosptial, Durban
  - Chris Hani Baragwanath Academic Hosptial, Soweto

IPD SHARING:
Plan to Share IPD: No